CLINICAL TRIAL: NCT00017537
Title: Phase IB Trial of Active Specific Immunotherapy With MVF-HER-2(628-647) and CRL1005 Copolymer Adjuvant in Patients With Metastatic Cancer
Brief Title: Vaccine Therapy in Treating Patients With Metastatic or Recurrent Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068700; UAB-0020; NCI-G01-1955
Record Dates: First submitted 2001-06-06; First posted 2004-01-08 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Gastric Cancer; Lung Cancer; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; adenocarcinoma of the stomach; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose #1 (Experimental): dose #1 administered
  Interventions: Biological: MVF-HER-2(628-647)-CRL 1005 vaccine
- Dose #2 (Experimental): dose #2 administered
  Interventions: Biological: MVF-HER-2(628-647)-CRL 1005 vaccine
- Dose #3 (Experimental): Dose #3 administered
  Interventions: Biological: MVF-HER-2(628-647)-CRL 1005 vaccine
- Dose #4 (Experimental): Dose #4 administered
  Interventions: Biological: MVF-HER-2(628-647)-CRL 1005 vaccine
- Dose #5 (Experimental): Administered dose #5
  Interventions: Biological: MVF-HER-2(628-647)-CRL 1005 vaccine

INTERVENTIONS:
Biological: MVF-HER-2(628-647)-CRL 1005 vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic or recurrent cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the optimum biologic dose of MVF-HER-2(628-647)-CRL 1005 vaccine that will induce anti-HER-2 antibody in patients with metastatic or recurrent cancer. II. Characterize the nature and severity of toxicity of this drug in these patients. III. Document any clinical responses to this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients receive MVF-HER-2(628-647)-CRL 1005 vaccine intramuscularly on days 1 and 29. Cohorts of 5 patients receive escalating doses of MVF-HER-2(627-647)-CRL 1005 vaccine until at least 2 of 5 patients experience dose-limiting toxicity. Patients are followed on days 43 and 57 and every 2 months for at least 1 year.

PROJECTED ACCRUAL: Approximately 5-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic and/or recurrent solid tumor, especially the following: Breast Ovarian Non-small cell lung cancer Gastric adenocarcinoma No standard therapy available No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL ALT less than 2 times upper limit of normal No hepatitis A, B, or C Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No serious cardiopulmonary disorder No congestive heart failure No symptomatic coronary artery disease No serious cardiac arrhythmia Pulmonary: No serious cardiopulmonary disorder No symptomatic chronic obstructive pulmonary disease Immunologic: Reactive to at least 1 of the following skin test antigens: Candida, mumps, Trichophyton, intermediate strength PPD, tetanus toxoid No concurrent disease requiring corticosteroids or other immunosuppressive drugs No autoimmune disease, including rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, or vasculitic syndrome No prior anaphylactic response to other vaccine No hypersensitivity to MVF-HER-2(628-647) Other: No active HIV No active infection requiring antibiotic therapy No serious medical disease Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: At least 4 weeks since prior cytotoxic chemotherapy and recovered Endocrine therapy: At least 4 weeks since prior hormonal therapy and recovered No concurrent corticosteroids Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: At least 4 weeks since prior surgery and recovered No prior splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Determine the optimum biologic dose of MVF-HER-2 (628-647)-CRL 1005 vaccine that will induce snit-HER-2 antibody in patients with metastatic or recurrent cancer | baseline to 1 year

SECONDARY OUTCOMES:
Characterize the nature and severity of toxicity of this drug in these patients. | baseline to 1 year
Document any clinical responses to this drug in these patients. | baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre L. Triozzi, MD, Study Chair — University of Alabama at Birmingham